CLINICAL TRIAL: NCT01570218
Title: Randomized Clinical Trial Testing Musicotherapy in the Reduction of Fatigue in Women With Breast or Gynecological Cancer Under Radiotherapy.
Brief Title: Musicotherapy in the Reduction of Fatigue in Women With Breast or Gynecological Cancer Under Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: Associaçao de Combate ao Cancer em Goias (Unknown)
Responsible Party: Principal Investigator, Ruffo Freitas-Junior, Professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RGM-02
Record Dates: First submitted 2012-03-17; First posted 2012-04-04 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer; Uterine Cancer; Ovarian Cancer
Keywords: breast cancer; gynecological cancer; radiotherapy; fatigue; musicotherapy
MeSH Terms: conditions — Breast Neoplasms; Uterine Neoplasms; Ovarian Neoplasms; Fatigue | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy (Experimental): Music therapy arm: Intervention with 10 sections of music therapy will be performed, twice a week, during 45 days.
  Interventions: Behavioral: Music therapy
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Music therapy — Music therapy arm: Intervention with 10 sections of music therapy will be performed, twice a week, during 45 days
  Other Names: musictherapy
  Arms: Music therapy

SUMMARY:
OBJETIVE: To study the influence of musicotherapy in reduction of fatigue related to cancer in patients with breast's or gynecology's cancer, during the radiotherapy treatment.

DETAILED DESCRIPTION:
METHODS: This is a randomized controled study (Control Group - CG e musicotherapy Group - MTG) wich values fatigue, life's quality, anxiety, depression by using evaluative instruments Functional Assessment of Cancer Therapy: Fatigue (FACT-F), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI) in three different moments (during first week of radiotherapy, in the intermediate phase's week and during the last week of radiotherapy) for patients of both groups. Women allocated in MTG, in addition to the scales described above, answered the musicotherapy Questionary (MQ), and the Subjective Impression of the Subject's Questionary in last meeting. Musicotherapy sessions were individual and lasted an average of 40 minutes. Music therapeutic techniques used were Musical Audition (MA) and Therapeutic Musical Audition (TMA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast and gynecological cancer with indication for radiotherapy
* Performance status 0,1

Exclusion Criteria:

* Hemoglobin < 10mg/dl
* Patients in psychotherapy during the study
* Use of antidepressants
* Patients presenting more than one cancer type

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Assess the influence of musicotherapy in the reduction of fatigue | 45 days
  To study the influence of musicotherapy in reduction of fatigue related to cancer in patients with breast or gynecological cancer, during the radiotherapy treatment.

SECONDARY OUTCOMES:
Assess the reduction of depression | 45 days
  To compare the levels of depression of patients with breast and gynecological cancer on radiotherapy, between the musicotherapy and the control group.
Asses the reduction of anxiety | 45 days
  To compare the levels of anxiety of patients with breast and gynecological cancer on radiotherapy, between the musicotherapy and the control group.
Assess the quality of life | 45 days
  To compare the levels of quality of life of patients with breast and gynecological cancer on radiotherapy, between the musicotherapy and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Ruffo Freitas-Junior, PhD, Study Chair — Universidade Federal de Goias; Tereza R Alcantara-Silva, Ms Mus, Principal Investigator — Universidade Federal de Goias
Locations (2):
- Brazil (2):
  - Goias Anticancer Association, Goiânia, Goiás
  - Hospital Araujo Jorge, Associacao de Combate ao Cancer em Goias, Goiânia, Goiás